CLINICAL TRIAL: NCT03326544
Title: Ultra-sound Guided Saphenous Nerve Block Versus Platelet Rich Plasma for Chronic Knee Joint Osteoarthritis
Brief Title: Saphenous Nerve Block Versus Platelet Rich Plasma for Chronic Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MS/17.07.80
Record Dates: First submitted 2017-10-26; First posted 2017-10-31 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Chronic Knee Joint Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saphenous nerve block group (Experimental): Patients will receive ultrasound-guided intervention treatment with a sub-sartorial approach for a saphenous nerve block with 8 mL of bupivacaine 0.5% plus dexamethasone 4 mg
  Interventions: Other: Saphenous nerve block group
- Platelet rich plasma group (Experimental): Patients will receive intra-articular ultrasound-guided injection of 5 mL of autologous Platelet rich plasma
  Interventions: Other: Platelet rich plasma group

INTERVENTIONS:
Other: Saphenous nerve block group — Patients will receive ultrasound-guided intervention treatment with a sub-sartorial approach for a saphenous nerve block with 8 mL of bupivacaine 0.5% plus dexamethasone 4 mg
  Arms: Saphenous nerve block group
Other: Platelet rich plasma group — Patients will receive intra-articular ultrasound-guided injection of 5 mL of autologous Platelet rich plasma
  Arms: Platelet rich plasma group

SUMMARY:
Knee osteoarthritis, as a progressive disease is one of the most common causes of pain, motor disorder and disability in the elderly. By increasing age, the cartilage is eroded and endures degenerative changes due to physiological and biomechanical changes as well as metabolic effects and trauma . Non-surgical interventions for pain control of knee osteoarthritis include weight loss, exercise, changes in daily activities, physiotherapy, nonsteroidal anti-inflammatory drugs (NSAIDs) and analgesics .However ,the intra-articular injection is recently recommended by many studies such as corticosteroids, hyaluronic acid, Growth hormone, dextrose ,and platelet rich plasma.

Intra-articular injection of platelets are activated and undergo degranulation, releasing a range of growth factors, including transforming growth factor beta (TGF-β), platelet-derived growth factor (PDGF), insulin-like growth factor, vascular endothelial growth factors, epidermal growth factors and basic fibroblast growth factor 2. These growth factors are thought to activate a variety of signaling pathways, which promote healing of bone and soft tissue.Also,some minimally invasive therapeutic options have been effective in pain relieve in KA, such as ultrasound-guided saphenous nerve block .

DETAILED DESCRIPTION:
The aim of this study is to compare the efficacy of ultrasound guided saphenous nerve block versus platelet rich plasma injection in the management of chronic pain in patients with knee OA. This study will be conducted to evaluate which modality is more effective.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are not competent to understand the study protocol
* Radiographic evidence of OA of knee of 2nd degree.
* Chronic pain for at least 6 months prior to study entry (day 0).
* Pain relief not achieved with conservative therapies during the last 6 months

Exclusion Criteria:

* Patient refusal.
* Bleeding disorders.
* Coagulation disorders.
* Local skin infection
* Current other problem in the affected extremity .
* Psychiatric disorders affecting co-operation of the patient .
* Previous chronic opioid use.
* Intra articular knee injection within previous three months.
* History of traumatic arthropathy.
* History of neuropathic arthropathy.
* Allergy or hypersensitivity to any of the study medication.
* Any condition that could interfere with the interpretation of the outcome assessments.
* Pregnancy
* Lactating women.
* low back pain due to central cause.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Pain scores | For 6 months after intervention
  The severity of pain will be assessed using a visual analog scale (VAS)

SECONDARY OUTCOMES:
Quality of life (QOL) | For 6 months after intervention
  is evaluated using the Western Ontario and MC Master universities (WOMAC) index of osteoarthritis

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospitals, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided